CLINICAL TRIAL: NCT00535210
Title: The Effects of a Group Exercise Program on Function in Spinal Cord Injury Rehabilitation: A Pilot Randomized Controlled Trial
Brief Title: The Effect of an Exercise Program on Physical Function After a Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unsuccessful recruiting patients, never got beyond pilot testing of patients
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Janice Eng, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H07-01073
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; exercise rehabilitation; inpatient; RCT; physical function
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other)
  Interventions: Behavioral: Cardiovascular training
- 2 (Other)
  Interventions: Behavioral: Balance training

INTERVENTIONS:
Behavioral: Cardiovascular training — The cardiovascular training group will receive their usual therapy plus 3 days of 30 minutes of exercise per week. This program will last for 6 weeks while the participant is in the hospital. The cardiovascular training program will include pushing and pulling on pulleys, wheeling over mats, punching a boxing bag, and using an arm ergometer. The balance training group will receive their usual therapy plus 3 days of 30 minutes of sitting balance activities. This program will last for 6 weeks while the participant is in the hospital.
  Arms: 1
Behavioral: Balance training — The balance training group will receive their usual therapy plus 3 days of 30 minutes of sitting balance activities. This program will last for 6 weeks while the participant is in the hospital. The balance training program will include sitting on mats - moving arm support from in front of the body to behind body, moving from sitting to lying and back up, and catching soft foam ball thrown directly to centre of chest and throwing it back.
  Arms: 2

SUMMARY:
This study would focus on adding a group exercise program to the usual therapy delivered in the hospital. We propose to design an exercise program that would be 30 minutes in length, 3 times per week. A medical doctor and physiotherapist would oversee the design and monitoring of the program.

We believe that this program will: 1) Increase the potential for better health, thus improving independence and quality of life; 2) Help people make the move from therapist run exercise to self management of exercise; 3) Engage the patient in the therapy process and place an expectation of active participation on the client; and 4) Promote physical activity as part of a healthy lifestyle.

DETAILED DESCRIPTION:
In total 30 participants admitted for spinal cord injury rehabilitation at GF Strong Rehabilitation Centre will be randomly assigned to either cardiovascular training group or balance training group. The cardiovascular training group will receive their usual therapy plus 3 days of 30 minutes of exercise per week. This program will last for 6 weeks while the participant is in the hospital. The cardiovascular training program will include pushing and pulling on pulleys, wheeling over mats, punching a boxing bag, and using an arm ergometer. The balance training group will receive their usual therapy plus 3 days of 30 minutes of sitting balance activities. This program will last for 6 weeks while the participant is in the hospital. The balance training program will include sitting on mats - moving arm support from in front of the body to behind body, moving from sitting to lying and back up, and catching soft foam ball thrown directly to centre of chest and throwing it back.

ELIGIBILITY:
Inclusion Criteria:

1. Sustained a traumatic spinal cord injury,
2. 16-50 years of age,
3. Able to push a manual wheelchair and arm ergometer,
4. Able to participate in exercise three times per week for 30 minutes,
5. Able to follow English instructions.

Exclusion Criteria:

1. Unstable cardiovascular status (congestive heart failure, uncontrolled hypertension, uncontrolled atrial fibrillation, or left ventricular failure),
2. Significant musculo-skeletal problems (e.g., rheumatoid arthritis) or neurological conditions (e.g., Parkinson's disease) due to conditions other than spinal cord injury,
3. Increased pain with exercise.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2007-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome is physical function. This outcome will be measured before and after the program. | 6 months

SECONDARY OUTCOMES:
Secondary outcomes include sitting balance and blood pressure in response to changes in position. Both these measures will be evaluated before and after the program. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Janice Eng, Ph.D, Principal Investigator — University of British Columbia; William Miller, Ph.D, Study Director — University of British Columbia; Andrei Krassioukov, Ph.D, Study Director — University of British Columbia; Chihya Hung, Study Chair — University of British Columbia; Amira Tawashy, Study Chair — University of British Columbia
Locations (1):
- GF Strong Rehab Research Lab, Vancouver, British Columbia, Canada